CLINICAL TRIAL: NCT05939206
Title: rTARUP (Robotic-assisted Transabdominal Retromuscular Umbilical Prosthetic Repair): Long-term Analysis of More Than 48 Months
Brief Title: rTARUP: Long-term Analysis
Acronym: rTARUP FU
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, MD, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: rTARUP FU
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Umbilical Hernia; TARUP; Robotic Abdominal Wall Surgery
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: rTARUP — robotic assisted transabdominal retromuscular umbilical prosthetic repair

SUMMARY:
The aim of the study is to assess the recurrence rate and potential long-term complications, at least 48 months, after a robotic assisted transabdominal retromuscular approach (rTARUP technique) for the repair of an umbilical hernia.

DETAILED DESCRIPTION:
The rTARUP technique (robotic assisted transabdominal retromuscular umbilical prosthetic repair) has been introduced in the latest years for the treatment of ventral/umbilical hernias. Short-term analyses have proven that this technique can be performed safely and without complications. The technique maintains the benefits of a traditional laparoscopic approach (smaller incision, faster recovery, shorter hospital stay) and obeys mesh complications related to intraperitoneal mesh placement (adhesions, pain due to mesh fixation). An initial evaluation was conducted at our center to assess recurrence and complications 1 year after the procedure in a patient group of 203 patients. We documented 3 patients with a recurrence of which 2 of them had a laparoscopic intra-peritoneal hernia repair to treat the recurrence. Due to Covid-19 restrictions a clinical follow-up was only possible in 73% of patients. Therefore, we believe that a longer follow-up period of at least 48 months after surgery is necessary and surgically relevant to analyze the primary (recurrence rate) and secondary (long-term complications) end points of the recently introduced rTARUP technique for the treatment of ventral/umbilical hernias.

Muysoms, F., et al., Robotic transabdominal retromuscular umbilical prosthetic hernia repair (TARUP): observational study on the operative time during the learning curve. Hernia, 2018. 22(6): p. 1101-1111.

Muysoms, F., et al., Observational study with one year follow-up on robotic assisted retro-rectus ventral hernia repair (RTARUP) with a self-fixating mesh. Br J Surg, 2021. 108(Suppl 8).

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent rTARUP procedure in the period September 2016 - December 2019
* Lateral approach to the retromuscular plane/lateral single docking
* Use of Progrip self-fixating mesh

Exclusion Criteria:

* Ventral hernia on the lateral side or combined hernia (lateral and medial)
* eTEP approach to the retromuscular plane
* Use of any other mesh than Progrip self-fixating mesh.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent rTARUP procedure in the period September 2016 - December 2019
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2023-04-22 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | After at least 48 months post-operative
  Hernia recurrence

SECONDARY OUTCOMES:
Long-term complications | After 48 months post-operative
  Long-term complications
Quality of Life Questionnaire | After 48 months post-operative
  Minimum score is 0, maximum score is 90. The higher the score, the worse the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided